CLINICAL TRIAL: NCT00703846
Title: A PHASE 4, OPEN-LABEL STUDY TO ASSESS THE LONG-TERM SAFETY OF EXTINA (KETOCONAZOLE) FOAM, 2% IN THE TREATMENT OF SEBORRHEIC DERMATITIS
Brief Title: STUDY TO ASSESS THE LONG-TERM SAFETY OF EXTINA (KETOCONAZOLE) FOAM, 2%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114568; NCT01337284 (obsolete NCT alias)
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Results first posted 2012-02-23 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Dermatitis, Seborrheic
Keywords: Phase 4; Seborrheic; Ketoconazole; Dermatitis
MeSH Terms: conditions — Dermatitis, Seborrheic; Dermatitis | interventions — Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KETOCONAZOLE (Other)
  Interventions: Drug: Ketoconazole

INTERVENTIONS:
Drug: Ketoconazole — Foam, 2%, Extina will be applied twice daily (morning and evening) to all seborrheic dermatitis lesions on the face, scalp, ears, neck, and chest. Study product should be applied at the first sign of a seborrheic dermatitis flare, and twice daily applications should continue until the area(s) has cleared. All symptom flares should be treated throughout the 12-month study period.

SUMMARY:
Extina (ketoconazole) Foam, 2% was approved for marketing in the United States (US) in June 2007. Extina foam is indicated for topical treatment of seborrheic dermatitis in immunocompetent patients 12 years of age and older. The approved dosing regimen is twice daily for 4 weeks. The treatment of recurrent seborrheic dermatitis demands a topical preparation that is safe for both short-term and chronic application. This study is being conducted in order to obtain long-term safety data on the use of Extina (ketoconazole) Foam, 2% in the treatment of seborrheic dermatitis.

DETAILED DESCRIPTION:
This is an open-label, multicenter, single-group study to assess the long-term safety of twice daily treatment with Extina (ketoconazole) Foam, 2% in subjects with seborrheic dermatitis.

The study subjects must have seborrheic dermatitis with an Investigator's Static Global Assessment (ISGA) of 2, 3, or 4 at baseline. In addition, subjects must have a discrete, evaluable target area of at least 0.5 cm2, with a score of 2, 3, or 4 for erythema and scaling.

All subjects will apply Extina (ketoconazole) Foam, 2% topically twice a day (morning and evening) to all seborrheic dermatitis lesions on the face, scalp, ears, neck, and chest. Study product should be applied at the first sign of a seborrheic dermatitis flare, and twice daily applications should continue until the area(s) has cleared. All symptom flares should be treated throughout the 12-month study period. Study visits will occur at baseline (day 1) and at weeks 4, 8, 16, 26, 39, and 52 (or early withdrawal). See the study flowchart (section 3) for the assessments to be performed at each visit. Primary Objective: To assess the long-term safety of Extina (ketoconazole) Foam, 2% in the treatment of seborrheic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following conditions or characteristics in order to be considered for study enrollment:

1. Capable of understanding and willing to provide signed and dated written voluntary informed consent before any protocol-specific procedures are performed. For subjects between the ages of 12 and 17 years, a parent or legal guardian must be capable of understanding and willing to sign informed consent and subject must be capable of understanding and willing to sign an adolescent assent.
2. Male or female subjects 12 years of age or older.
3. Able to complete the study and to comply with study instructions.
4. Female subjects of childbearing potential must have a negative pregnancy test. Sexually active women of childbearing potential participating in the study must use a medically acceptable form of contraception (which includes oral contraception, injectable or implantable methods, or intrauterine devices). Barrier methods of contraception are not acceptable. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant. Abstinence is considered an appropriate barrier control method.
5. Seborrheic dermatitis on the face, scalp, ears, neck, or chest with an ISGA of 2, 3, or 4 at baseline
6. Subjects must have a discrete, evaluable target area of at least 0.5 cm2, with a score of 2, 3, or 4 for erythema and scaling on the Seborrheic Dermatitis Grading Scale

Exclusion Criteria:

Subjects with any of the following conditions or characteristics will be excluded from study enrollment:

1. Use of systemic antifungal agents, corticosteroids or other immunosuppressive therapies, or systemic retinoids within 4 weeks prior to the baseline visit.
2. Use of topical antifungal therapy, corticosteroid therapy, or calcineurin inhibitors to the face, scalp, ears, neck, or chest within 2 weeks prior to the baseline visit.
3. Use of any investigational drugs within 8 weeks prior to the baseline visit, or subjects who are scheduled to receive an investigative drug other than the study product during the period of the study.
4. History of known or suspected intolerance to any of the ingredients of the study product.
5. Female subjects who are pregnant, trying to become pregnant, or lactating.
6. Any clinically relevant abnormal vital signs or findings on the physical examination.
7. A clinically relevant history of abuse of alcohol or other drugs.
8. Any major illness within 30 days prior to the baseline visit.
9. Subjects with any clinically significant condition which would, in the opinion of the investigator, compromise the subject's participation in the study.
10. Subjects who are immunocompromised.
11. Considered unable or unlikely to attend the necessary visits.
12. Employees of Stiefel Laboratories or a contract research organization involved in the study, or an immediate family member (partner, offspring, parents, siblings, or sibling's offspring) of an employee.
13. Currently using any medication, which in the opinion of the investigator may affect the evaluation of the study product or place the subject at undue risk.
14. Only one subject per household may be entered into the study. These inclusion and exclusion criteria will be strictly adhered to throughout the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2008-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Draelos ZD, Feldman SR, Butners V, Alio Saenz AB. Long-term safety of ketoconazole foam, 2% in the treatment of seborrheic dermatitis: results of a phase IV, open-label study. J Drugs Dermatol. 2013 Jan;12(1):e1-6. PMID 23377341
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 114568 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114568 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114568 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114568 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114568 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114568 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114568 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Extina (Ketoconazole) 2%: Extina (ketoconazole) Foam, 2% was topically applied twice a day (morning and evening [BD]) to all seborrheic dermatitis lesions on the face, scalp, ears, neck, and chest until the areas were cleared. The maximum treatment period was 12 months.
Period: Overall Study
Arm/Group | Extina (Ketoconazole) 2%
Started | 500
Completed | 363
Not Completed | 137
Not completed — Adverse Event | 8
Not completed — Lost to Follow-up | 55
Not completed — Lack of Efficacy | 15
Not completed — Noncompliance with Study Treatment | 2
Not completed — Withdrawal by Subject | 40
Not completed — Death | 1
Not completed — Other | 14
Not completed — Did Not Receive Study Drug | 2

BASELINE CHARACTERISTICS:
Groups:
- Extina (Ketoconazole) 2%: Extina (ketoconazole) Foam, 2% was topically applied at the first sign of a seborrheic dermatitis flare, and twice a day (morning and evening [BD]) to all seborrheic dermatitis lesions on the face, scalp, ears, neck, and chest until the areas were cleared. All symptom flares were treated throughout the 12-month study period.
Arm/Group | Extina (Ketoconazole) 2%
Number analyzed (Participants) | 498
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline Characteristics were collected in the Safety Analysis Set Population, comprised of all participants who were randomized and received at least one dose of study drug. Two participants did not receive any study treatment and are thus not included in this population.
  Years | 47.2 (17.4)
Gender [Count of Participants; unit: Participants]
  Female | 239
  Male | 259
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 20
  Asian | 8
  Black | 108
  Multiracial | 14
  Native Hawaiian or Other Pacific Islander | 2
  White | 346

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, which does not necessarily have a causal relationship with the treatment. For a list of all adverse events occurring at or above a frequency threshold of 5% during the course of the study, see the table entitled "Other (Non-Serious) Adverse Events."
Time Frame: From baseline through 52 weeks
Population: Safety Analysis Set: all participants who had used the study product at least once
Measure: Number; unit: participants
Groups:
- Extina (Ketoconazole) 2%: Extina (ketoconazole) Foam, 2% was topically applied at the first sign of a seborrheic dermatitis flare, and BD to all seborrheic dermatitis lesions on the face, scalp, ears, neck, and chest until the areas were cleared. All symptom flares were treated throughout the 12-month study period.
Arm/Group | Extina (Ketoconazole) 2%
Number analyzed (Participants) | 498
participants | 282

2. Secondary Outcome: Mean Change From Baseline in Skin Assessments for Erythema at Weeks 4, 8, 16, 26, 39, and 52 (or Early Termination)
Description: Mean change from baseline was calculated as the Week 4, 8, 16, 26, 39, and 52 (or early termination) value minus the baseline value. The grading scale for erythema ranges from 0 to 4; 0=Normal skin without erythema; may have residual hyper/hypopigmentation; 1=Faint erythema; may have residual hyper/hypopigmentation; 2=Light red erythema; may have residual hyper/hypopigmentation; 3=Moderate red coloration; 4=Dusky to deep red coloration. Erythema was defined as redness of the skin caused by increased blood circulation in the capillaries found in the deeper layers of the skin.
Time Frame: Baseline and Weeks 4, 8, 16, 26, 39, and 52 (or early termination)
Population: Safety Analysis Set. Participants withdrew from the study as the study progressed, and data were missing for some participants. There were no imputation methods used for missing data for any analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Extina (Ketoconazole) 2%
Number analyzed (Participants) | 451
units on a scale
  Week 4, n=451 | -2 (1.02)
  Week 8, n=436 | -2 (0.98)
  Week 16, n=405 | -2 (0.93)
  Week 26, n=381 | -2 (0.91)
  Week 39, n=370 | -2 (0.95)
  Week 52 (or Early Termination), n=420 | -2 (1.03)

3. Secondary Outcome: Mean Change From Baseline in Skin Assessments for Scaling at Weeks 4, 8, 16, 26, 39, and 52 (or Early Termination)
Description: Mean change from baseline in skin assessments for scaling was calculated as the Week 4, 8, 16, 26, 39, and 52 (or Early Termination) value minus the baseline value. The grading scale for scaling ranges from 0 to 4; 0=Normal skin with rare fine scale; 1=Minimal: occasional fine scales over less than 10% of the lesions; 2=Mild: fine scales predominate; 3=Moderate: coarse scales predominate; 4=Severe: thick tenacious scales predominate. Scaling of skin is the loss of the outer layer of the epidermis in large, scale-like flakes.
Time Frame: Baseline and Weeks 4, 8, 16, 26, 39, and 52 (or early termination)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Extina (Ketoconazole) 2%
Number analyzed (Participants) | 451
units on a scale
  Week 4, n=451 | -2 (1.03)
  Week 8, n=436 | -2 (1.00)
  Week 16, n=405 | -2 (0.93)
  Week 26, n=381 | -2 (0.98)
  Week 39, n=370 | -2 (1.03)
  Week 52 (or Early Termination), n=420 | -2 (1.07)

4. Secondary Outcome: Mean Change From Baseline in Skin Assessments for Pruritus at Weeks 4, 8, 16, 26, 39, and 52 (or Early Termination)
Description: Mean change from baseline was calculated as the Week 4, 8, 16, 26, 39, and 52 (or Early Termination) value minus the baseline value. The grading scale for pruritis ranges from 0 to 4; 0=No itching; 1=Minimal: rarely aware of itching; 2=Mild: only aware of itching at times; only present when relaxing; not present when focused on other activities; 3=Moderate: often aware of itching; annoying; sometimes disturbs sleep and daytime activities; 4=Severe: constant itching; distressing; frequent sleep disturbance; interferes with activities. Pruritus is defined as an itching/scratching sensation.
Time Frame: Baseline and Weeks 4, 8, 16, 26, 39, and 52 (or early termination)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Extina (Ketoconazole) 2%
Number analyzed (Participants) | 451
units on a scale
  Week 4, n=451 | -2 (1.22)
  Week 8, n=436 | -2 (1.13)
  Week 16, n=405 | -2 (1.11)
  Week 26, n=381 | -2 (1.13)
  Week 39, n=370 | -2 (1.07)
  Week 52 (or Early Termination), n=420 | -2 (1.13)

5. Secondary Outcome: Mean Change From Baseline in Investigator's Static Global Assessment (ISGA) at Weeks 4, 8, 16, 26, 39, and 52 (or Early Termination)
Description: This seborrhoeic dermatitis-specific ISGA scale (range=0-4) is used to assess skin condition severity without considering changes over time ("static"). 0=clear, except for minor residual discoloration; 1-4=majority of lesions have average scaling/erythema scores of 1-4, respectively. 1=almost clear, occasional fine scale, faint erythema/barely perceptible plaque thickness; 2= mild, fine scale with light coloration/mild plaque elevation; 3=moderate, coarse scale with moderate red coloration/moderate plaque thickness; 4=severe, thick tenacious scale with deep coloration/severe plaque thickness.
Time Frame: Baseline and Weeks 4, 8, 16, 26, 39, and 52 (or early termination)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Extina (Ketoconazole) 2%
Number analyzed (Participants) | 451
units on a scale
  Week 4, n=451 | -1 (0.94)
  Week 8, n=436 | -2 (0.91)
  Week 16, n=405 | -2 (0.88)
  Week 26, n=381 | -2 (0.94)
  Week 39, n=370 | -2 (0.98)
  Week 52 (or Early Termination), n=420 | -2 (1.04)

6. Secondary Outcome: Median Number of Flares
Description: The median number of flares for all participants was calculated based on data self-reported in diaries that participants kept during the study. A flare is defined as a clinical diagnosis and presentation of seborrheic dermatitis that shows as an erythematous, thin, scaly patch with a greasy sandpaper texture that varies depending on disease severity. Flares are commonly seen on the scalp, nasal folds, eyebrows, glabella, upper eyelids, retroauricular/external ear canal, and midchest areas.
Time Frame: From baseline through 52 weeks
Population: Safety Analysis Set
Measure: Median (Full Range); unit: flares
Arm/Group | Extina (Ketoconazole) 2%
Number analyzed (Participants) | 498
flares | 7 [1 to 68]

7. Secondary Outcome: Median Number of Flare Days
Description: The median number of flare days for all participants was calculated based on data self-reported in diaries that participants kept during the study. The median number of flares for all participants was calculated based on data self-reported in diaries that participants kept during the study. A flare day is defined as a day on which flare signs and symptoms for seborrheic dermatitis (erythema, scaling, and pruritus of the target area) occurred.
Time Frame: From baseline through 52 weeks
Population: Safety Analysis Set
Measure: Median (Full Range); unit: flare days
Arm/Group | Extina (Ketoconazole) 2%
Number analyzed (Participants) | 498
flare days | 109 [1 to 365]

8. Secondary Outcome: Mean Change From Baseline for the Global Score of the Participant-completed Skindex-29 Quality of Life Questionnaire at Week 52 (or Early Termination)
Description: Skindex-29 is a 3-component (symptomatic, emotional, and functional) self-administered questionnaire (comprised of 30 questions) used to comprehensively measure the complex effects of skin diseases on a participant's quality of life. Participants were asked to answer questions based on a 5-point scale concerning their feelings over the past 4 weeks about the skin condition that has bothered them the most: 1, never; 2, rarely; 3, sometimes; 4, often; 5, all the time. The Global Score is the sum of the 30 question scores; total score ranges from 30 to 150.
Time Frame: Baseline and Week 52 (or Early Termination)
Population: Safety Analysis Set. Participants who submitted incomplete questionnaires (missing values) were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Extina (Ketoconazole) 2%
Number analyzed (Participants) | 412
units on a scale | -11 (17.90)

9. Secondary Outcome: Mean Change From Baseline for the Symptomatic Score of the Participant-completed Skindex-29 Quality of Life Questionnaire at Week 52 (or Early Termination)
Description: Skindex-29 is a 3-component (symptomatic, emotional, and functional) self-administered questionnaire (comprised of 30 questions) used to comprehensively measure the complex effects of skin diseases on a participant's quality of life. For the symptomatic component, participants were asked to answer 7 questions based on a 5-point scale concerning their feelings over the past 4 weeks about the skin condition that has bothered them the most: 1, never; 2, rarely; 3, sometimes; 4, often; 5, all the time. The Symptomatic Score is the sum of the 7 question scores; total score ranges from 7 to 35.
Time Frame: Baseline and Week 52 (or Early Termination)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Extina (Ketoconazole) 2%
Number analyzed (Participants) | 412
units on a scale | -3 (5.13)

10. Secondary Outcome: Mean Change From Baseline for the Emotional Score of the Participant-completed Skindex-29 Quality of Life Questionnaire at Week 52 (or Early Termination)
Description: Skindex-29 is a 3-component (symptomatic, emotional, and functional) self-administered questionnaire (comprised of 30 questions) used to comprehensively measure the complex effects of skin diseases on a participant's quality of life. For the emotional component, participants were asked to answer 10 questions based on a 5-point scale concerning their feelings over the past 4 weeks about the skin condition that has bothered them the most: 1, never; 2, rarely; 3, sometimes; 4, often; 5, all the time. The Emotional Score is the sum of the 10 question scores; total score ranges from 10 to 50.
Time Frame: Baseline and Week 52 (or Early Termination)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Extina (Ketoconazole) 2%
Number analyzed (Participants) | 412
units on a scale | -5 (7.68)

11. Secondary Outcome: Mean Change From Baseline for the Functional Score of the Participant-completed Skindex-29 Quality of Life Questionnaire at Week 52 (or Early Termination)
Description: Skindex-29 is a 3-component (symptomatic, emotional, and functional) self-administered questionnaire (comprised of 30 questions) used to comprehensively measure the complex effects of skin diseases on a participant's quality of life. For the functional component, participants were asked to answer 15 questions based on a 5-point scale concerning their feelings over the past 4 weeks about the skin condition that has bothered them the most: 1, never; 2, rarely; 3, sometimes; 4, often; 5, all the time. The Functional Score is the sum of the 12 question scores; total score ranges from 15 to 75.
Time Frame: Baseline and Week 52 (or Early Termination)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Extina (Ketoconazole) 2%
Number analyzed (Participants) | 412
units on a scale | -4 (8.72)

ADVERSE EVENTS:
Arm/Group | Extina (Ketoconazole) 2%
Serious Adverse Events (participants affected / at risk) | 16/498
Other Adverse Events (participants affected / at risk) | 140/498
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Extina (Ketoconazole) 2% (N=498)
Coronary artery disease (Cardiac disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Oesophageal rupture (Gastrointestinal disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Breast cancer metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Psychotic disorder (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Extina (Ketoconazole) 2% (N=498)
Application site irritation (General disorders) | 38
Nasopharyngitis (Infections and infestations) | 41
Upper respiratory tract infection (Infections and infestations) | 29
Headache (Nervous system disorders) | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.